CLINICAL TRIAL: NCT01281735
Title: INTERNATIONAL STUDY of Chronic Myeloid Leukaemia (CML) Treatment and Outcomes in Children and Adolescents
Brief Title: International Chronic Myeloid Leukemia Pediatric Study
Acronym: ICMLPed
Status: Recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Collaborators: CIC Inserm 1402 (Unknown); University of Milano Bicocca (Other); University Medical Center Groningen (Other); University of Liege (Other); Imperial College London (Other); University Hospital Dresden (Other); International BFM Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: CIC1402; 2010-023359-27 (EudraCT Number)
Record Dates: First submitted 2011-01-14; First posted 2011-01-24 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Chronic Myeloid Leukemia
Keywords: treatment outcome; side effects; Protein Kinase Inhibitors; pediatrics
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to describe and characterize CML in a large pediatric cohort of patients.

DETAILED DESCRIPTION:
International study of CML in children and adolescents

1. Rational and objectives 1.1 Rational: Chronic myeloid leukaemia (CML) is a malignant disease of the hematopoietic system characterized by the presence a reciprocal translocation between chromosome 9 and 22. CML is a very rare disease in children and adolescents, accounting for 2% to 3% of leukemias in this age range, with an annual incidence of 1 case per million children (1,2,3). A recent report of the French National Registry of childhood leukemia and lymphoma revealed an incidence of 0.6 case per million children under 15 years of age between 1990 and 1999 in France. Characteristics of CML seem to differ in this age range compared with adults (5). In Europe, very few children and adolescents with CML is included in national trials nor are they recorded in regional or national registries. A European CML-Registry was established to improve the knowledge concerning this disease but only patients aged 18 years and over are registered. In Europe, a national registry was recently set up in UK to collect prospectively data in patients less than 15 years of age with CML. However, limited information is available concerning the epidemiology and the characteristics of CML in childhood.

   There are currently two main treatment options in children with CML. The first option is allogeneic hematopoietic transplantation which is a potentially curative therapy in children with a suitable donor. Transplantation with a matched unrelated donor resulted in an overall survival rate of 66% at 3 years in children with CML in first chronic phase (6). A 5-year overall survival rate of 73 % was reported in those transplanted with a matched sibling donor (7). The second option is treatment with imatinib mesylate, an orally administered antityrosine kinase. Imatinib mesylate is well tolerated and cytogenetic and molecular remissions can be achieved in a significant percentage of children with CML (8, 9). However, the ability of imatinib mesylate to cure the disease remains unknown.

   In adults with CML, Sokal and Hasford reported 2 distinct staging systems able to distinguish patient groups with different survival. These scoring systems were determined in cohorts of patients including adults and children, but the data of the younger patients were not analysed separately. Moreover, the Sokal score was determined in patients treated with busulfan or hydroxyurea and the Hasford score in patients receiving IFN therapy. Identification of prognosis factors and determination of a prognostic scoring system in children and adolescents with CML are essential to optimize individual treatment strategy in this age group. All these points justify the need for an international network to better describe this rare disease in children and adolescents and to optimize individual treatment strategy.

   1.2 Objectives.

   The main objectives of the study are the followings:
   * To describe the characteristics of CML in a large cohort of patients less than 18 years of age
   * To describe the treatment policies.
   * To identify prognostic factors in this age-group
   * To determine prognostic scoring systems in this population in order to optimize individual treatment choices.
   * To determine side effects and long term effects of treatments, mainly the tyrosine kinase inhibitor effect, on growth and development of a pediatric population
2. Population. All patients less than 18 years of age with newly diagnosed Philadelphia positive and/or bcr-abl positive CML are eligible whatever the phase of the disease, the type of treatment and the enrollment or not in a clinical study.

   However their data will be collected only if requirements concerning ethics and policy agreement are fulfilled (see section 9)
3. Method The study is strictly observational. Retrospective and prospective data will be collected from patient flow charts and/or existing databases.

   A steering committee (SC) including A Biondi, E De Bont, MF Dresse, J de la Fuente, M Suttorp, J Guilhot and F Millot will promote the international study of CML in children and adolescents. The SC will include representatives of each country involved in the study. The SC will agree on policy, support its implementation, initiate research, and raise public awareness about the study by presentations and publications.A scientific committee (SciC) will be set up. By laws regarding data property,analysis and publication will be decided by the scientific committee and the steering committee. For each objective of the study, there will be a working party (WP),which will be open to all interested participants in the study.Data will be provided by clinicians and biologists involved in pediatric haematology.The data base of the study will be set up in the Clinical Investigation Center(CIC INSERM 802)of the University Hospital of Poitiers(France)which will be the International Central Data Center(ICDC) of the study in charge of and centralizing the data. Sophie Zin Ka Yeu will be the responsible for the monitoring,E Ducasse for data base management and J Guilhot for the statistical analysis. The study is international.A National Coordinating Center and a leader will be identified in each participating country. The National Coordinating Center will be in charge of collecting data for his country. Each leader of the National Coordinating Center will be in charge of registering the patients and sending the data to the ICDC (CIC INSERM 802, Poitiers, France). To avoid double entry, the location of the medical center where the CML of the patient was diagnosed will be recorded in the case report form. Moreover, notification of new cases may be cross checked by national coordinators with their own national registry when available (for example with the Registre national des hémopathies malignes de l'enfant in France).
4. Origin and type of data:

   Data will include:
   * Identification number
   * Demographic data
   * Date of birth
   * Sex
   * Medical data Ethnicity will be collected because of variation in terms of clinical characteristics (height for example) and pharmacokinetic of medication of the different groups of children potentially involved. Identifying biological results will not be collected.

   The ICDC will collect only data which is strictly anonymized by the national coordinating centers. Patients will be identified by a code including 2 to 3 letters for the country and 4 digits for the patient number (ex: FR/0001 for the first registered Patient in France). No initial of patients will be used. As country coordinator for France, F Millot will also collect initials of French patients in order to avoid double registration. These initials will not be computerized. The international ID number will be immediately provided.
5. Circulation of the data The data is centralized in the ICDC of the study. The ICDC is located in the Clinical Research Investigation Center of the University Hospital of Poitiers (France).

   Retrospective data:the data will be collected in a one step procedure. Prospective data:The data will be collected using a two step procedures.
   1. Notification of the cases:

      New cases will be notified by physicians and biologists involved in pediatric hematology to their National Coordinating Center; at regular intervals these cases will then be referred by this coordinating center to the ICDC.
   2. Full data collection:

   The data will be collected from the clinical chart of the patients. The complete data will be send to each National Coordinating Center and then centralized at regular intervals subsequently in the ICDC. Follow up will be required twice a year. For each case of CML, a yet to be fixed sum of money will be transferred from the ICDC to the National Coordinating Center at notification of the case and when complete data transfer will be performed.

   To avoid extra work, data already computerized will be accepted if it fulfilled the requirements of ethics, confidentiality and partnership rules as mentioned in paragraph 7.

   When available agreement between parties, data may come from case report form of patients included in clinical studies or other Registries. Data will be sent by regular mail, fax or electronic file by the national coordinators to the ARC of the study at the ICDC. Data received by mail will be transferred by copy using disks (CD-Rom or external disk) to the data-manager and destroyed from the computer with mail box. Data will be entered in a Microsoft ACCESS database in the ICDC. Data base will be implemented in a PC (I) (Windows) located in a room dedicated for the purpose of the work. A second PC (II) in the same place will be used for duplication, backup, quality control and analysis of the data. None of these 2 PCs will offer connections such as Internet, or Intranet. The use of an electronic case Report form (e-CRF) is not planned. A secure access building and rooms of the ICDC is organized; specific password and login for the computers are used. At regular interval a secure storage of the data will be performed and located in the secure IDCD room organized for this purpose. Access to the data will be restricted to the coordinator of the study, the ARC, the data manager, the biostatistician, and Health Authorities, if needed.
6. Study duration and organization The expected start date is August 1, 2009. The planned study duration is about 5 years. Study prolongation will depend on the funding linked to the effective participation of the centres in the study.
7. Analysis of the data Data will be analysed using mainly SAS software (SAS institute, CARY, NC, USA). Final analyses will be provided within 5 years from start of the study. Analysis will be mainly descriptive. Date of inclusion in the study is defined as the date of reception of the notification of case by the ICDC. For the purpose of descriptive analysis, all parameters will be analysed at regular intervals: number of registered cases, baseline characteristics, follow-up and outcome variables. Categorical data will be presented with frequency, percentage and 95 % confidence interval. Quantitative variable will be presented with median and range, mean and standard deviation when relevant. Survival data and issue to events (time to response or side-effects, loss and duration of response…); will be analysed by the Kaplan Meier and competing risks methods. For prognosis factors identification, exploratory analyses will be performed as appropriate. The final statistical plan will be validated by the steering committee and the scientific committee.

   Reports will be provided every 6 months and by the end of the study by the ARC, the data manager, the biostatistician and Dr F. Millot, coordinator of the study. These reports will be sent to the national coordinators and to the participants. Results could be presented in Workshops, meetings and could be published with the agreement of the steering and scientific committees. All reports and publications will remain anonymous.
8. Number of Patients :

   A proximately 100 to 150 patients per year are expected. As the number of cases of children and adolescent with CML being low, no strict calculation was made. The objective is to collect a maximum of cases to improve the power of the study.
9. Ethical Considerations The children, according to their age, and their parents will be informed about the study and its procedures, according to the European policy regarding collection and transfer data for research purpose. Informed consent (parents and, when possible, children) will have to be provided.

Anonymized data will be collected and presented in this study. Rules will be in accordance with the Principles and Guideline of the European Community concerning clinical studies and data collection and the French Law "Informatique, fichiers et liberté" (January 6, 1978, updated.It is the responsibility of each national coordinator to provide insurance concerning the participation of the members of his groups according these rules and the local rules required by his own country.

ELIGIBILITY:
Inclusion Criteria:

* patients less than 18 years of age
* diagnosed Philadelphia positive and/or BCR-ABL positive Chronic Myeloid Leukemia (CML) all phases

Exclusion Criteria:

* patients more than 18 years of age at diagnosis of CML

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients less than 18 years of age with newly diagnosed Philadelphia positive and/or bcr-abl positive CML are eligible whatever the phase of the disease, the type of treatment and the enrollment or not in a clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2011-01; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic MILLOT, MD, Principal Investigator — Poitiers University Hospital
Locations (20):
- Women's and children's Hospital, North Adelaide, South Australia, Australia
- St. Anna Children's Cancer Research Institute and St. Anna Children's Hospital, Vienna, Austria
- Belarussian Reseach Center for Pediatric Oncology and hematology (BRCPOH), Minsk, Belarus
- University Hospital of Ghent, Ghent, Belgium
- Instituto de Oncologia Pediatrica, São Paulo, Brazil
- Hospital Roberto Del Rio, Santiago, Chile
- Prince of Wales Hospital, Hong Kong, China
- Children's Hospital Zagreb, Zagreb, Croatia
- Charles University Motol, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- Clinical Investigation Center CIC 1402, Poitiers, France
- University Hospital Dresden, Dresden, Germany
- Agia Sophia Children's Hospital, Athens, Greece
- Keio University School of Medicine, Tokyo, Japan
- Saint George Hospital University Medical Centre, Beirut, Lebanon
- Dutch Childhood Oncology Group, Princess Maxima Center for pediatric oncology, Utrecht, Netherlands
- Wroclaw Medical University Department, Wroclaw, Poland
- University Children's Hospital, Bratislava, Slovakia
- Officina Proyectos SEHOP, Palma de Mallorca, Spain
- Uludag University, Medical Faculty, Görükle, Turkey (Türkiye)

REFERENCES:
- [Derived] Millot F, De Keizer J, Metzler M, Kalwak K, Gunes AM, De Moerloose B, Luesink M, Honrubia AM, Sedlacek P, Yajima J, Ampatzidou M, Dworzak M, Lausen B, Borisevich M, Li CK, Kolenova A, Jakovljevic G, Farah R, Durocher L, Baruchel A, Suttorp M. Children with chronic phase chronic myeloid leukemia: characteristics and outcomes from the International Registry of Childhood CML. Haematologica. 2025 Oct 23. doi: 10.3324/haematol.2025.288283. Online ahead of print. PMID 41126742
- [Derived] Meyran D, Petit A, Guilhot J, Suttorp M, Sedlacek P, De Bont E, Li CK, Kalwak K, Lausen B, Culic S, de Moerloose B, Biondi A, Millot F. Lymphoblastic predominance of blastic phase in children with chronic myeloid leukaemia treated with imatinib: A report from the I-CML-Ped Study. Eur J Cancer. 2020 Sep;137:224-234. doi: 10.1016/j.ejca.2020.06.024. Epub 2020 Aug 13. PMID 32799036
- [Derived] Millot F, Maledon N, Guilhot J, Gunes AM, Kalwak K, Suttorp M. Favourable outcome of de novo advanced phases of childhood chronic myeloid leukaemia. Eur J Cancer. 2019 Jul;115:17-23. doi: 10.1016/j.ejca.2019.03.020. Epub 2019 May 10. PMID 31082688
- [Derived] Millot F, Guilhot J, Suttorp M, Gunes AM, Sedlacek P, De Bont E, Li CK, Kalwak K, Lausen B, Culic S, Dworzak M, Kaiserova E, De Moerloose B, Roula F, Biondi A, Baruchel A. Prognostic discrimination based on the EUTOS long-term survival score within the International Registry for Chronic Myeloid Leukemia in children and adolescents. Haematologica. 2017 Oct;102(10):1704-1708. doi: 10.3324/haematol.2017.170035. Epub 2017 Aug 24. PMID 28838993